CLINICAL TRIAL: NCT05801419
Title: Nicotine Influence on Vascularization and Retinal Metabolism Following Electronic Cigarette Use
Brief Title: Nicotine Influence on the Retina Following the Use of Electronic Cigarette
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Casanova (Industry)
Responsible Party: Sponsor-Investigator, Christian Casanova, Professor, Zilia Inc.
Organization: Zilia Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZRC07
Record Dates: First submitted 2022-09-26; First posted 2023-04-06 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Electronic Cigarette Use; Retina; Change
MeSH Terms: conditions — Vaping | interventions — Electronic Nicotine Delivery Systems; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Baseline, post e-cigarette without nicotine and post e-cigarette with nicotine (Experimental): Pattern visual event-related potential (ERP) and pattern electroretinogram (pERG) on right eye (non-dilated pupil), followed by eye fundus tissue oximetry on left eye (dilated pupil), followed by optical coherence tomography angiography (OCT-A) on left eye (dilated pupil).
  Interventions: Device: RETI-port/scan 21; Device: Zilia Ocular; Device: OCT-A; Combination Product: Electronic cigarette without nicotine; Combination Product: Electronic cigarette with nicotine

INTERVENTIONS:
Device: RETI-port/scan 21 — Pattern visual event-related potential and pattern electroretinogram on right eye (non-dilated pupil) at baseline, post e-cigarette vaping without nicotine and post e-cigarette vaping with nicotine.
Device: Zilia Ocular — Eye fundus tissue oximetry measure on left eye (dilated pupil) at baseline, post e-cigarette vaping without nicotine and post e-cigarette vaping with nicotine.
Device: OCT-A — Optical coherence tomography angiography measure on left eye (dilated pupil) at baseline, post e-cigarette vaping without nicotine and post e-cigarette vaping with nicotine.
Combination Product: Electronic cigarette without nicotine — Vaping using an e-cigarette paired with an e-cigarette liquid vial without nicotine. Inhaling through the mouth and exhaling through the nose ten times. Inhalations must last 5 seconds and the participant has 5 minutes to do the 10 inhalations.
Combination Product: Electronic cigarette with nicotine — Vaping using an e-cigarette paired with an e-cigarette liquid vial with nicotine. Inhaling through the mouth and exhaling through the nose ten times. Inhalations must last 5 seconds and the participant has 5 minutes to do the 10 inhalations.

SUMMARY:
The marketing of electronic cigarettes (e-cigarettes) in 2003 was initially intended to present a healthier alternative to smokers. Subsequently, it became an extremely widespread fashion phenomenon, especially among young people. It thus contributes to attracting new consumers thanks to its modern and technological presentation, combined with a panoply of captivating fragrances.

In 2014, the FDA still does not recognize this practice as a substitute for smoking intended to limit it, and several recent studies have demonstrated the potential harmful effects of e-cigarettes on health. Indeed, the latter also have pulmonary effects reminiscent of those of the original cigarette, namely breathing difficulties or even lung inflammation.

In addition, a potential impact on the vascular system has recently been highlighted by the use of these e-cigarettes. Thus, their components can lead to vascular changes in the reactivity of blood vessels, an increase in blood pressure or even endothelial dysfunction and vascular and cerebral oxidative stress.

The aim of this study is to detect these phenomena at the level of the retinal circulation, window of the central nervous system, in order to be able to confirm the acute vascular impacts of the use of an e-cigarette. In addition, the vascular and metabolic impacts due to the potential toxicity of the other components of these e-cigarettes could be investigated. Finally, the comparison between patients who are smokers and occasional smokers will provide a better understanding of the different acute and chronic effects of nicotine.

ELIGIBILITY:
Inclusion Criteria:

* Subject between 18 and 40 years old.
* The subject must be a regular smoker (more than 1 cigarette per day for 2 years) OR be an occasional smoker (between 1 and 15 cigarettes in his life).
* The subject must be able to sign a free and informed consent, and to follow the instructions.
* Complete visual examination within the last 5 years.

Exclusion Criteria:

* Narrow iridocorneal angles.
* Inadequate or contraindicated pupil dilation.
* Insufficient visual fixation.
* Ametropia greater than -6 and +6 δ.
* Known hypersensitivity or allergy to any component of the ophthalmic formulation used, including benzalkonium chloride (preservative) and components of the vaping liquid.
* Eye trauma or eye surgery in the last 6 months.
* Evidence of present or recent infection or inflammation in both eyes.
* The use of ocular or systemic medication 30 days prior to the study.
* Presence of ocular pathology (corneal oedema, severe keratoconjunctivitis sicca, advanced cataract, retinopathy, glaucoma).
* Systemic disease (uncontrolled diabetes, myasthenia gravis...) or pulmonary, cardiac, hepatic, renal, endocrine problems.
* History of epilepsy and psychiatric: schizophrenia, bipolarity, anxiety, depression.
* Being pregnant or breastfeeding.
* History of alcohol abuse.
* History of drug or psychotropic use.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Change in retinal electric activity between baseline, after use of e-cigarette without nicotine and after use of e-cigarette with nicotine | At baseline, approximately 13 after baseline and after approximately 28 minutes after baseline
  Assessed with pattern visual event-related potential (ERP)
Change in visual cortex response between baseline, after use of e-cigarette without nicotine and after use of e-cigarette with nicotine | At baseline, approximately 13 after baseline and after approximately 28 minutes after baseline
  Assessed with pattern electroretinogram (pERG)
Change in eye fundus tissue oxygen saturation between baseline, after use of e-cigarette without nicotine and after use of e-cigarette with nicotine | At baseline, approximately 13 after baseline and after approximately 28 minutes after baseline
  Assessed with eye fundus tissue oximetry
Change in retinal capillaries density between between baseline, after use of e-cigarette without nicotine and after use of e-cigarette with nicotine | At baseline, approximately 13 after baseline and after approximately 28 minutes after baseline
  Assessed with optical coherence tomography angiography (OCT-A)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Casanova, PhD, Principal Investigator — École d'optométrie de l'Université de Montréal
Locations (1):
- École d'optométrie de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No